CLINICAL TRIAL: NCT04040803
Title: Characterizing the Application of Transcranial Alternating Current Stimulation and Transcranial Random Noise Stimulation Over Human Pharyngeal Motor Cortex
Brief Title: tACS and tRNS Studies on Brain Control of Swallowing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Prof Shaheen Hamdy PhD FRCP, Principal Investigator, University of Manchester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-5932-10164
Record Dates: First submitted 2019-04-25; First posted 2019-08-01 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Dysphagia; Swallowing Disorder
Keywords: transcranial alternating current stimulation; transcranial random noise stimulation; frequency; full spectrum
MeSH Terms: conditions — Deglutition Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: All people studied will have each of the five treatments separately over different days in random order.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 10 Hz tACS (Experimental): Stimulation will be applied at 10 Hz tACS with an intensity of 1.5 mA (peak to peak), a fade in/out of 10 s and a duration of 10min.
  10 Hz tACS will be performed over the pharyngeal cortex region and contralateral supraorbital region.
  Interventions: Device: Transcranial alternating current stimulation (tACS) and transcranial random noise stimulation (tRNS)
- 20 Hz tACS (Experimental): Stimulation will be applied at 20 Hz tACS with an intensity of 1.5 mA (peak to peak), a fade in/out of 10 s and a duration of 10min.
  20 Hz tACS will be performed over the pharyngeal cortex region and contralateral supraorbital region.
  Interventions: Device: Transcranial alternating current stimulation (tACS) and transcranial random noise stimulation (tRNS)
- 70Hz tACS (Experimental): Stimulation will be applied at 70 Hz tACS with an intensity of 1.5 mA (peak to peak), a fade in/out of 10 s and a duration of 10min.
  70 Hz tACS will be performed over the pharyngeal cortex region and contralateral supraorbital region.
  Interventions: Device: Transcranial alternating current stimulation (tACS) and transcranial random noise stimulation (tRNS)
- 0.1-640Hz tRNS (Experimental): Stimulation will be applied at 0.1-640Hz tRNS with an intensity of 1.5 mA (peak to peak), a fade in/out of 10 s and a duration of 10min.
  0.1-640Hz tRNS will be performed over the pharyngeal cortex region and contralateral supraorbital region.
  Interventions: Device: Transcranial alternating current stimulation (tACS) and transcranial random noise stimulation (tRNS)
- Sham (Sham Comparator): Stimulation will be performed only for 10 s before the fade out, with 20 Hz tACS and an intensity of 1.5 mA (peak to peak).
  Sham condition will be applied over pseudo-stimulation of pharyngeal cortex region and contralateral supraorbital region.
  Interventions: Device: Transcranial alternating current stimulation (tACS) and transcranial random noise stimulation (tRNS)

INTERVENTIONS:
Device: Transcranial alternating current stimulation (tACS) and transcranial random noise stimulation (tRNS) — Transcranial alternating current stimulation (tACS) and transcranial random noise stimulation (tRNS) are two (CE marked medical devices) new, non-invasive (over the scalp) brain stimulation (NIBS) techniques. Both tACS and tRNS deliver a weak current continuously across the brain using pads placed over the scalp, which has been shown safe and well-tolerated by healthy adults and patients. These two techniques are able to softly alter physiological function within the brain. tACS can influence the brainwaves which have been demonstrated to play important roles in movement, sensation, and thinking functions. tACS and tRNS have been investigated for several years and have been shown to be safe, well tolerated and produce beneficial results in hand movement, hearing, and working memory.

SUMMARY:
Transcranial alternating current stimulation (tACS) and transcranial random noise stimulation (tRNS) are two (CE marked medical devices) new, non-invasive (over the scalp) brain stimulation (NIBS) techniques. Both tACS and tRNS deliver a weak current continuously across the brain using pads placed over the scalp, which has been shown safe and well-tolerated by healthy adults and patients. These two techniques are able to softly alter physiological function within the brain. tACS can influence the brainwaves which have been demonstrated to play important roles in movement, sensation, and thinking functions. tACS and tRNS have been investigated for several years and have been shown to be safe, well tolerated and produce beneficial results in hand movement, hearing, and working memory.

Swallowing problems are life-threatening symptom among patients with brain impairments and elderly people. Until now, there are no studies investigating whether tACS and tRNS can have a beneficial effect on swallowing function in human. Our aim is to examine the effects of different strengths of tACS and tRNS to determine the best approach for brain stimulation that controls swallowing action, before using these techniques in patients with (neurological) swallowing disorders.

Participants: Healthy adults who are aged 18 years old or above with no medical complications or significant past medical history will be recruited in the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults who are aged 18 years old or above with no medical complications or significant past medical history

Exclusion Criteria:

* a history of epilepsy
* cardiac pacemaker
* previous brain surgery
* previous swallowing problems
* risk of potential pregnancy
* metal in the head or eyes
* use of medication that acts on the central nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Changes of pharyngeal motor evoked potential amplitudes (PMEPs) | These cortical excitability measurements will be recorded at baseline, followed by immediately after intervention, then every 15 minutes up to 120 minutes afterwards.
  Cortical excitability of the pharyngeal motor cortices are being assessed as the primary endpoints. Therefore, the changes in EMG pharyngeal motor evoked potential amplitudes (PMEPs) following the intervention applied to pharyngeal motor cortex are being collected.

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Hamdy, MD,PhD, Principal Investigator — GI-sciences, Salford Royal NHS Foundation Trust, University of Manchester
Locations (1):
- Upper G.I laboratory, Salford Royal Hospital, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The Gastrointestinal Sciences research team at the University of Manchester will have access to participants' identifiable information, but it will be anonymized as soon as participants are enrolled in this study. Representatives from the University of Manchester and regulatory authorities will have access to the anonymised data if required for auditing and monitoring process. However, participants' anonymised consent form, contact details, and data collected for this study will be retained for 5 years.

REFERENCES:
- [Background] Antal A, Herrmann CS. Transcranial Alternating Current and Random Noise Stimulation: Possible Mechanisms. Neural Plast. 2016;2016:3616807. doi: 10.1155/2016/3616807. Epub 2016 May 3. PMID 27242932
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Herrmann CS, Munk MH, Engel AK. Cognitive functions of gamma-band activity: memory match and utilization. Trends Cogn Sci. 2004 Aug;8(8):347-55. doi: 10.1016/j.tics.2004.06.006. PMID 15335461
- [Background] Engel AK, Fries P, Singer W. Dynamic predictions: oscillations and synchrony in top-down processing. Nat Rev Neurosci. 2001 Oct;2(10):704-16. doi: 10.1038/35094565. PMID 11584308
- [Background] Pollok B, Boysen AC, Krause V. The effect of transcranial alternating current stimulation (tACS) at alpha and beta frequency on motor learning. Behav Brain Res. 2015 Oct 15;293:234-40. doi: 10.1016/j.bbr.2015.07.049. Epub 2015 Jul 28. PMID 26225845
- [Background] Wach C, Krause V, Moliadze V, Paulus W, Schnitzler A, Pollok B. Effects of 10 Hz and 20 Hz transcranial alternating current stimulation (tACS) on motor functions and motor cortical excitability. Behav Brain Res. 2013 Mar 15;241:1-6. doi: 10.1016/j.bbr.2012.11.038. Epub 2012 Dec 3. PMID 23219965
- [Background] Jausovec N, Jausovec K. Increasing working memory capacity with theta transcranial alternating current stimulation (tACS). Biol Psychol. 2014 Feb;96:42-7. doi: 10.1016/j.biopsycho.2013.11.006. Epub 2013 Nov 27. PMID 24291565
- [Background] Riecke L, Formisano E, Herrmann CS, Sack AT. 4-Hz Transcranial Alternating Current Stimulation Phase Modulates Hearing. Brain Stimul. 2015 Jul-Aug;8(4):777-83. doi: 10.1016/j.brs.2015.04.004. Epub 2015 Apr 24. PMID 25981160
- [Background] Clave P, Shaker R. Dysphagia: current reality and scope of the problem. Nat Rev Gastroenterol Hepatol. 2015 May;12(5):259-70. doi: 10.1038/nrgastro.2015.49. Epub 2015 Apr 7. PMID 25850008
- [Result] Jefferson S, Mistry S, Singh S, Rothwell J, Hamdy S. Characterizing the application of transcranial direct current stimulation in human pharyngeal motor cortex. Am J Physiol Gastrointest Liver Physiol. 2009 Dec;297(6):G1035-40. doi: 10.1152/ajpgi.00294.2009. Epub 2009 Oct 8. PMID 19815630
- [Result] Moliadze V, Atalay D, Antal A, Paulus W. Close to threshold transcranial electrical stimulation preferentially activates inhibitory networks before switching to excitation with higher intensities. Brain Stimul. 2012 Oct;5(4):505-11. doi: 10.1016/j.brs.2011.11.004. Epub 2012 Feb 22. PMID 22445135
- [Result] Uhlhaas PJ, Singer W. Abnormal neural oscillations and synchrony in schizophrenia. Nat Rev Neurosci. 2010 Feb;11(2):100-13. doi: 10.1038/nrn2774. PMID 20087360
- [Result] Moisa M, Polania R, Grueschow M, Ruff CC. Brain Network Mechanisms Underlying Motor Enhancement by Transcranial Entrainment of Gamma Oscillations. J Neurosci. 2016 Nov 23;36(47):12053-12065. doi: 10.1523/JNEUROSCI.2044-16.2016. PMID 27881788
- [Result] Fertonani A, Pirulli C, Miniussi C. Random noise stimulation improves neuroplasticity in perceptual learning. J Neurosci. 2011 Oct 26;31(43):15416-23. doi: 10.1523/JNEUROSCI.2002-11.2011. PMID 22031888
- [Result] Rjosk V, Kaminski E, Hoff M, Gundlach C, Villringer A, Sehm B, Ragert P. Transcranial Alternating Current Stimulation at Beta Frequency: Lack of Immediate Effects on Excitation and Interhemispheric Inhibition of the Human Motor Cortex. Front Hum Neurosci. 2016 Nov 3;10:560. doi: 10.3389/fnhum.2016.00560. eCollection 2016. PMID 27857687
- [Result] Terney D, Chaieb L, Moliadze V, Antal A, Paulus W. Increasing human brain excitability by transcranial high-frequency random noise stimulation. J Neurosci. 2008 Dec 24;28(52):14147-55. doi: 10.1523/JNEUROSCI.4248-08.2008. PMID 19109497